CLINICAL TRIAL: NCT01254279
Title: Multicentre, Single-arm, Open Label Clinical Trial Intended to Provide Early Access to Cabazitaxel in Patients With Metastatic Hormone Refractory Prostate Cancer Previously Treated With a Docetaxel-containing Regimen and to Document Safety of Cabazitaxel in These Patients
Brief Title: Early Access to Cabazitaxel in Patients With Metastatic Hormone Refractory Prostate Cancer Previously Treated With a Docetaxel-containing Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABAZ_C_05331; 2010-021128-92 (EudraCT Number); U1111-1115-2476 (Other: UTN)
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — cabazitaxel

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel 25 mg/m² intravenously every 3 weeks, in combination with oral prednisone or prednisolone 10 mg daily
  Interventions: Drug: CABAZITAXEL

INTERVENTIONS:
Drug: CABAZITAXEL — Pharmaceutical form: Concentrate For Solution For Infusion Route of administration: Intravenous

SUMMARY:
The purpose of this study is to allow patients similar to that evaluated in the TROPIC trial (NCT00417079), and Investigators access to cabazitaxel for the management of metastatic Hormone Refractory Prostate Cancer (mHRPC) in those patients who have progressed during or after docetaxel and to document the overall safety of cabazitaxel in these patients.

Please note that in each country, patient recruitment will end when cabazitaxel becomes commercially available.

ELIGIBILITY:
Inclusion criteria:

* Metastatic Hormone Refractory Prostate Cancer (mHRPC) previously treated with a docetaxel-containing regimen
* Disease Progression during or after docetaxel-containing regimen for mHRPC
* Surgical or medical castration
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0-2
* Life-expectancy ≥3 months
* Adequate bone marrow, liver, and renal function: Neutrophils> 1500 /mm3; Hemoglobin > 10 g/dL; Platelets > 100 x109/L; Bilirubin < ULN; SGOT (AST) < 1.5xULN; SGPT (ALT) < 1.5xULN; Creatinine < 1.5xULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance < 60 mL/min should be excluded.

Exclusion criteria:

* Prior radiotherapy to ≥ 40% of bone marrow
* Prior radionuclide therapy (samarium-153, strontium-89, P-32…)
* Prior surgery, radiation, chemotherapy, or other anti-cancer therapy within 4 weeks prior to enrollment
* Active grade ≥2 peripheral neuropathy
* Active grade ≥2 stomatitis
* Active infection requiring systemic antibiotic or anti-fungal medication
* Active cancer (other than mHRPC) including prior malignancy from which the patient has been disease-free for ≤5 years (except superficial basal cell skin cancer)
* Known brain or leptomeningeal involvement
* History of severe hypersensitivity reaction (≥grade 3) to docetaxel
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
* History of severe hypersensitivity reaction (≥grade 3) or intolerance to prednisone or prednisolone
* Uncontrolled severe illness or medical condition (including uncontrolled cardiac arrhythmias, angina pectoris, hypertension or diabetes mellitus). History of congestive heart failure (NYHA III or IV) or myocardial infarction within last 6 months is also not allowed.
* Concurrent or planned treatment with potent inhibitors or inducers of cytochrome P450 3A4/5
* Participation in a clinical trial with any investigational drug
* Patient with reproductive potential not implementing accepted and effective method of contraception

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To provide early access to cabazitaxel in patients with metastatic hormone refractory prostate cancer previously treated with a docetaxel-containing regimen | Up to 30 weeks

SECONDARY OUTCOMES:
To document safety of cabazitaxel in these patients | Up to 35 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (165):
- Australia (22):
  - Investigational Site Number 036004, Box Hill
  - Investigational Site Number 036020, Campbelltown
  - Investigational Site Number 036001, Camperdown
  - Investigational Site Number 036002, Camperdown
  - Investigational Site Number 036011, Douglas
  - Investigational Site Number 036019, Nambour
  - Investigational Site Number 036023, North Adelaide
  - Investigational Site Number 036008, Parkville
  - Investigational Site Number 036005, Perth
  - Investigational Site Number 036003, Port Macquarie
  - Investigational Site Number 036025, Randwick
  - Investigational Site Number 036009, South Brisbane
  - Investigational Site Number 036022, South Brisbane
  - Investigational Site Number 036017, Southport
  - Investigational Site Number 036012, St Leonards
  - Investigational Site Number 036010, Sydney
  - Investigational Site Number 036013, Sydney
  - Investigational Site Number 036014, Sydney
  - Investigational Site Number 036016, Tweed Heads
  - Investigational Site Number 036024, Wendouree
  - Investigational Site Number 036007, Westmead
  - Investigational Site Number 036015, Wodonga
- Austria (4):
  - Investigational Site Number 040-004, Linz
  - Investigational Site Number 040-005, Salzburg
  - Investigational Site Number 040-002, Vienna
  - Investigational Site Number 040-003, Vienna
- Belgium (7):
  - Investigational Site Number 056002, Bruges
  - Investigational Site Number 056007, Brussels
  - Investigational Site Number 056003, Haine-Saint-Paul
  - Investigational Site Number 056005, Liège
  - Investigational Site Number 056004, Ottignies
  - Investigational Site Number 056001, Roeselare
  - Investigational Site Number 056006, Tournai
- Bosnia and Herzegovina (3):
  - Investigational Site Number 070003, Banja Luka
  - Investigational Site Number 070001, Sarajevo
  - Investigational Site Number 070002, Zenica
- Bulgaria (4):
  - Investigational Site Number 100004, Plovdiv
  - Investigational Site Number 100001, Sofia
  - Investigational Site Number 100003, Sofia
  - Investigational Site Number 100002, Sofia
- Canada (10):
  - Investigational Site Number 124012, Kitchener
  - Investigational Site Number 124009, Laval
  - Investigational Site Number 124004, London
  - Investigational Site Number 124007, Moncton
  - Investigational Site Number 124001, Montreal
  - Investigational Site Number 124011, Montreal
  - Investigational Site Number 124010, Québec
  - Investigational Site Number 124003, Toronto
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124006, Winnipeg
- Investigational Site Number 191-001, Zagreb, Croatia
- Investigational Site Number 203001, Brno, Czechia
- Denmark (3):
  - Investigational Site Number 208-001, Cph Ø
  - Investigational Site Number 208-002, Herlev
  - Investigational Site Number 208-003, Odense
- Finland (2):
  - Investigational Site Number 246002, Helsinki
  - Investigational Site Number 246001, Seinäjoki
- Hungary (4):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348002, Szolnok
  - Investigational Site Number 348003, Szombathely
  - Investigational Site Number 348004, Veszprém
- India (5):
  - Investigational Site Number 356004, Chennai
  - Investigational Site Number 356006, Gūrgaon
  - Investigational Site Number 356001, New Delhi
  - Investigational Site Number 356002, New Delhi
  - Investigational Site Number 356005, Trivandrum
- Ireland (4):
  - Investigational Site Number 372004, Cork
  - Investigational Site Number 372001, Dublin
  - Investigational Site Number 372002, Dublin
  - Investigational Site Number 372003, Dublin
- Italy (25):
  - Investigational Site Number 380-001, Arezzo
  - Investigational Site Number 380-011, Aviano
  - Investigational Site Number 380-025, Bari
  - Investigational Site Number 380-007, Bergamo
  - Investigational Site Number 380-015, Bologna
  - Investigational Site Number 380-021, Fano
  - Investigational Site Number 380-012, Florence
  - Investigational Site Number 380-003, Genova
  - Investigational Site Number 380-005, Genova
  - Investigational Site Number 380-014, Lecce
  - Investigational Site Number 380-023, Messina
  - Investigational Site Number 380-018, Milan
  - Investigational Site Number 380-022, Milan
  - Investigational Site Number 380-006, Napoli
  - Investigational Site Number 380-010, Napoli
  - Investigational Site Number 380-027, Napoli
  - Investigational Site Number 380-004, Orbassano
  - Investigational Site Number 380-017, Padua
  - Investigational Site Number 380-002, Parma
  - Investigational Site Number 380-009, Roma
  - Investigational Site Number 380-008, Roma
  - Investigational Site Number 380-024, Rozzano
  - Investigational Site Number 380-020, San Giovanni Rotondo
  - Investigational Site Number 380-013, Sassari
  - Investigational Site Number 380-016, Taormina
- Kazakhstan (2):
  - Investigational Site Number 398001, Almaty
  - Investigational Site Number 398003, Shymkent
- Investigational Site Number 442001, Niedercorn, Luxembourg
- Malaysia (3):
  - Investigational Site Number 458002, George Town
  - Investigational Site Number 458001, Kuala Lumpur
  - Investigational Site Number 458003, Kuching
- Mexico (4):
  - Investigational Site Number 484002, Durango
  - Investigational Site Number 484006, Irapuato
  - Investigational Site Number 484005, Toluca
  - Investigational Site Number 484001, Zapopan
- Investigational Site Number 608001, Manila, Philippines
- Investigational Site Number 616-001, Gdansk, Poland
- Portugal (5):
  - Investigational Site Number 620002, Coimbra
  - Investigational Site Number 620003, Lisbon
  - Investigational Site Number 620004, Lisbon
  - Investigational Site Number 620001, Porto
  - Investigational Site Number 620005, Setúbal
- Romania (3):
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642002, Cluj-Napoca
  - Investigational Site Number 642003, Timișoara
- Serbia (2):
  - Investigational Site Number 688001, Belgrade
  - Investigational Site Number 688002, Belgrade
- Singapore (2):
  - Investigational Site Number 702002, Singapore
  - Investigational Site Number 702001, Singapore
- Slovakia (2):
  - Investigational Site Number 703001, Bratislava
  - Investigational Site Number 703002, Košice
- Spain (25):
  - Investigational Site Number 724002, A Coruña
  - Investigational Site Number 724018, Barcelona
  - Investigational Site Number 724019, Barcelona
  - Investigational Site Number 724023, Castellon
  - Investigational Site Number 724020, Córdoba
  - Investigational Site Number 724025, Elche
  - Investigational Site Number 724017, Granada
  - Investigational Site Number 724006, Guadalajara
  - Investigational Site Number 724011, L'Hospitalet de Llobregat
  - Investigational Site Number 724010, León
  - Investigational Site Number 724003, Madrid
  - Investigational Site Number 724012, Madrid
  - Investigational Site Number 724007, Madrid
  - Investigational Site Number 724008, Manresa
  - Investigational Site Number 724021, Málaga
  - Investigational Site Number 724009, Oviedo
  - Investigational Site Number 724022, Pamplona
  - Investigational Site Number 724005, San Cristóbal de La Laguna - Santa Cruz de Tenerife
  - Investigational Site Number 724016, Santander
  - Investigational Site Number 724015, Santiago de Compostela
  - Investigational Site Number 724024, Seville
  - Investigational Site Number 724004, Terrassa
  - Investigational Site Number 724013, Valencia
  - Investigational Site Number 724014, Valencia
  - Investigational Site Number 724001, Zaragoza
- Sweden (2):
  - Investigational Site Number 752-002, Umeå
  - Investigational Site Number 752-001, Uppsala
- Taiwan (5):
  - Investigational Site Number 005, Kaohsiung Hsien,
  - Investigational Site Number 004, Taichung
  - Investigational Site Number 002, Taipei
  - Investigational Site Number 003, Taipei
  - Investigational Site Number 001, Tao Yuan Hsien
- United Kingdom (12):
  - Investigational Site Number 826011, Birmingham
  - Investigational Site Number 826002, Bristol
  - Investigational Site Number 826003, Glasgow
  - Investigational Site Number 826013, Leeds
  - Investigational Site Number 826009, London
  - Investigational Site Number 826012, Manchester
  - Investigational Site Number 826004, Metropolitan Borough of Wirral
  - Investigational Site Number 826005, Nottingham
  - Investigational Site Number 826008, Preston
  - Investigational Site Number 826001, Sutton
  - Investigational Site Number 826007, Torquay
  - Investigational Site Number 826006, Whitechurch

REFERENCES:
- [Derived] Bahl A, Masson S, Malik Z, Birtle AJ, Sundar S, Jones RJ, James ND, Mason MD, Kumar S, Bottomley D, Lydon A, Chowdhury S, Wylie J, de Bono JS. Final quality of life and safety data for patients with metastatic castration-resistant prostate cancer treated with cabazitaxel in the UK Early Access Programme (EAP) (NCT01254279). BJU Int. 2015 Dec;116(6):880-7. doi: 10.1111/bju.13069. Epub 2015 Jun 16. PMID 25639506
- [Derived] Castellano D, Anton Aparicio LM, Esteban E, Sanchez-Hernandez A, Germa JR, Batista N, Maroto P, Perez-Valderrama B, Luque R, Mendez-Vidal MJ; cabazitaxel EAP study. Cabazitaxel for metastatic castration-resistant prostate cancer: safety data from the Spanish expanded access program. Expert Opin Drug Saf. 2014 Sep;13(9):1165-73. doi: 10.1517/14740338.2014.939583. Epub 2014 Jul 7. PMID 25001524